CLINICAL TRIAL: NCT01430897
Title: Right Ventricular Hypertrophy After Atrial Switch Operation and Its Role in a Systemic RV: Normal Adaptation Process or Risk Factor? A Cardiovascular Magnetic Resonance Study
Brief Title: Right Ventricular Hypertrophy After Atrial Switch and Cardiovascular Magnetic Resonance (CMR) Findings
Status: Completed | Type: Observational
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Matthias Grothoff, M.D., Consultant Radiology, University of Leipzig
Other Study IDs: 261-11-22082011
Record Dates: First submitted 2011-09-05; First posted 2011-09-08 (Estimated); Last update posted 2011-09-08 (Estimated); Status verified 2011-09

CONDITIONS: Right Ventricular Hypertrophy; d-TGA
Keywords: d-TGA; dextro Transposition of the great arteries; systemic right ventricle; right ventricular failure; Atrial switch procedure
MeSH Terms: conditions — Hypertrophy, Right Ventricular; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Systemic RV hypertrophy and impaired systolic function occur after atrial switch (AS) in d-transposition of the great arteries (d-TGA). Echocardiography has limitation in the assessment of the right ventricle (RV).

In this study the investigators sought to evaluate systemic RV myocardial mass and function after AS for d-TGA and to analyze the role of excessive hypertrophy for ventricular function under special consideration of the interventricular septal (IVS) movement.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility criteria were an AS operation in childhood for correction of d-TGA and the absence of associated hemodynamically significant heart defects.

Exclusion Criteria:

* Exclusion criteria were usual CMR contraindications such as ferromagnetic metallic implants.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Thirty-seven consecutive patients who came to regular outpatient visits at our tertiary care institution were referred to CMR.
  Patient parameters were compared to a control group of 25 healthy age matched volunteers.
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2007-04; Primary Completion 2011-04 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Gutberlet, MD, Study Chair — University pf Leipzig - Heart Center
Locations (1):
- University of Leipzig - Heart Center, Leipzig, Germany

REFERENCES:
- [Result] Hornung TS, Kilner PJ, Davlouros PA, Grothues F, Li W, Gatzoulis MA. Excessive right ventricular hypertrophic response in adults with the mustard procedure for transposition of the great arteries. Am J Cardiol. 2002 Oct 1;90(7):800-3. doi: 10.1016/s0002-9149(02)02619-x. No abstract available. PMID 12356407